CLINICAL TRIAL: NCT01797432
Title: Safety and Efficacy of Combined Restylane and Triamcinolone Acetonide Injections for the Treatment of Alopecia Areata
Brief Title: Combined Restylane and Triamcinolone Acetonide Injections for the Treatment of Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0907M69801
Record Dates: First submitted 2012-07-06; First posted 2013-02-22 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combined IL Kenalog and Restylane (Experimental): Injection of Intralesional Triamcinolone Acetonide 10 mg/mL (Kenalog-10) on whole scalp and Restylane on half of scalp
  Interventions: Drug: Intralesional Triamcinolone Acetonide 10 mg/mL (Kenalog-10); Device: Restylane

INTERVENTIONS:
Drug: Intralesional Triamcinolone Acetonide 10 mg/mL (Kenalog-10) — Intralesional injections of 4mLs Triamcinolone Acetonide 10 mg/mL (Kenalog-10) on the whole scalp
  Other Names: Kenalog-10
Device: Restylane — Intralesional injections of 2mLs of Restylane on one side of the scalp

SUMMARY:
The investigators hypothesize that Restylane® could serve as a repair matrix which also maintains IL triamcinolone acetonide concentrations at higher levels for a longer period of time in the skin, giving a more sustained local anti-inflammatory effect and thus, arresting the AA process and promoting hair regrowth. Furthermore, the combination of Restylane® with IL triamcinolone acetonide injections may prevent a common side effect, atrophy. With the prevention of scalp atrophy and the preservation of higher concentrations of triamcinolone acetonide for longer periods of time, patients may see a better clinical response for a longer period of time. Quality of life may improve as the number of clinic visits decreases as would the number of IL corticosteroid injections.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18 and greater.
2. Alopecia areata diagnosis in the last two years with extensive scalp involvement, between 74% and 99%, alopecia areata must involve the left and right hemispheres of the scalp.
3. Willing to abstain from use of over the counter products and prescription products, other than study medications, which may promote hair growth.
4. Willing to abstain from the use of non-steroidal anti-inflammatory medications, aspirin, St. Johns Wart, and high doses of Vitamin E supplementation.
5. Subjects are capable of giving informed consent.
6. Willing to adhere to protocol, including scalp examinations and photography.

Exclusion Criteria:

1. Allergy or intolerance to Restylane® or hyaluronate preparations
2. Allergy or intolerance to triamcinolone acetonide, 10 mg/cc.
3. Underlying disease that might be adversely affected by Restylane® or triamcinolone (ex. patients with bleeding disorders).
4. Immunosuppressed patients (history of transplantation, cancer, chemotherapy, splenectomy, HIV).
5. Pregnant or lactating female.
6. Application of topical immunomodulatory or immunosuppressive agent in the preceding 6 weeks.
7. Systemic administration of corticosteroid or other systemic treatment (i.e. prednisone) that has immunomodulatory or other immunosuppressive mechanism of action, in the preceding 8 weeks.
8. Clinical evidence of secondary skin infection (i.e., folliculitis).
9. Other inflammatory or infectious skin disease that might interfere with evaluations during the study.
10. Investigational medications within the past 30 days.
11. Patients with susceptibility to keloid formation.
12. Severe allergies manifested by a history of anaphylaxis, or history or presence of multiple severe allergies
13. Patients with allergies to gram positive bacterial proteins
14. Unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota - Department of Dermatology
Locations (1):
- University of Minnesota Department of Dermatology, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combined IL Kenalog and Restylane
Started | 14
Completed | 10
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — lived too far from study site | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combined IL Kenalog and Restylane
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.43 (18.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Alopecia Areata Half Head Severity Score (AAHHSS) at 12 Weeks Compared to Baseline
Description: The primary endpoint of evaluating the efficacy of administration of IL triamcinolone acetonide 10 mg/cc and Restylane® in the management of AA is the alopecia areata half head severity score (AAHHSS) comparing week 12 with baseline hair loss. Four discreet areas of the scalp are examined. The percent of terminal hair loss in each area is measured by visual estimation. Those percent figures are multiplied by the total area on one half of the scalp represented by the four respective areas. 1) Left parietal scalp (18% of area), right parietal scalp (18% of area), frontal scalp (40% of area), and occipital scalp (24% of area). Scores range from 0 to 50, with higher scores indicating more hair loss.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined IL Kenalog and Restylane
Number analyzed (Participants) | 10
score on a scale | -17.75 (23.36)

2. Secondary Outcome: Number of Adverse Events Reported by Subjects
Description: To assess the safety of IL triamcinolone acetonide 10 mg/cc and Restylane® in the management of AA.
Time Frame: 12 weeks
Measure: Number; unit: adverse events
Arm/Group | Combined IL Kenalog and Restylane
Number analyzed (Participants) | 14
adverse events | 25

ADVERSE EVENTS:
Arm/Group | Combined IL Kenalog and Restylane
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined IL Kenalog and Restylane (N=14)
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Shingles (Infections and infestations) | 1 (1)
Bladder Infection (Renal and urinary disorders) | 1 (1)
Migraine Headache (General disorders) | 1 (1)
Cold Sore (Immune system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain at Injection Site (Skin and subcutaneous tissue disorders) | 1 (1)
Irregular Menstrual Cycle (Reproductive system and breast disorders) | 1 (1)
Cold/flu (Infections and infestations) | 1 (1)
Headache (General disorders) | 1 (1)
Difficulty Concentrating (General disorders) | 1 (1)
Traveler's Diarrhea (Gastrointestinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2)
Hives (Immune system disorders) | 1 (1)
Bump on Head (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-04-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT01797432/Prot_SAP_000.pdf
  • Informed Consent Form (2014-11-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT01797432/ICF_001.pdf